CLINICAL TRIAL: NCT03101631
Title: Exploratory Study of Frailty Evaluation in Elderly Population With Cancer
Brief Title: Frailty Evaluation in Elderly Population With Cancer
Acronym: ELDERLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Javier Gallego Plazas, PhD, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ELDERLY V 1.0 20DEC2012
Record Dates: First submitted 2017-03-17; First posted 2017-04-05 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Fragility; Cancer
Keywords: Elderly population with cancer; Toxicity risk; Mortality risk; Frailty conditions in elderly population; Chemotherapy in elderly population
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Cases and Contols Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CASE ARM (Experimental): This is a three cohorts arm with intervention (CGA):
  * Nutritional Assessment: Mini Nutritional Assessment (MNA)
  * Functional Assessment: Get up and Go, Activities of Daily Living (ADL), Instrumental Activities of Daily Living (IADL), Karnofsky Scale, Walking one Block, Number of Falls in last 6 months and Hearing Loss.
  * Cognitive Assessment: Mini-Mental State Examination (MMSE-30)
  * Psychological status: Geriatric Depression Scale (GDS)
  * Social Support: Medical Outcomes Study Social Support Survey (MOS-SSS)
  * Comorbidity and Severity of Comorbidities: Charlson Comorbidity Index and Adult Comorbidity Evaluation (ACE-27)
  * Age
  * Haemoglobin
  * Creatinine Clearance (CrCl)
  * Presence of Geriatric Syndromes
  Interventions: Diagnostic Test: Comprehensive Geriatric Assessment (CGA)
- CONTROL ARM (No Intervention): This is a three cohorts arm with no intervention

INTERVENTIONS:
Diagnostic Test: Comprehensive Geriatric Assessment (CGA) — CGA includes a set of evaluations to determine therapeutic decision based on mortality risk, toxicity risk and frailty group. Evaluations includes:
  * Nutritional Assessment: Mini Nutritional Assessment (MNA)
  * Functional Assessment: Get up and Go, Activities of Daily Living (ADL), Instrumental Activities of Daily Living (IADL), Karnofsky Scale, Walking one Block, Number of Falls in last 6 months and Hearing Loss.
  * Cognitive Assessment: Mini-Mental State Examination (MMSE-30)
  * Psychological status: Geriatric Depression Scale (GDS)
  * Social Support: Medical Outcomes Study Social Support Survey (MOS-SSS)
  * Comorbidity and Severity of Comorbidities: Charlson Comorbidity Index and Adult Comorbidity Evaluation (ACE-27)
  * Age
  * Haemoglobin
  * CrCl
  * Presence of geriatric syndromes
  Other Names: Frailty Evaluation
  Arms: CASE ARM

SUMMARY:
The Comprehensive Geriatric Assessment (CGA) is, still today, barely established in the standard practice. Although the different scientific societies recommend a CGA in elderly population affected with cancer at first visit, the evidence regarding its transcendence is limited. On the other hand, the components of this evaluation and the translation of their findings in changes in the clinical practice are not stablished. This project intends to implement a CGA in a group of patients to compare this group with an historical cohort that reflects the standard practice, to evaluate the differences between both approaches. The study also evaluate the feasibility and utility of this CGA. All these questions aims to support the hypothesis that CGA impacts on the cancer treatment for elderly population affected with cancer.

DETAILED DESCRIPTION:
This study compares two groups of elderly patients affected with stage IV non-small lung cancer (NSCLC), stage III colon cancer and stage IV colorectal cancer (CRC): a prospective experimental cohort and an historic control cohort. The sample size is 60 patients, 30 prospective and 30 retrospective. Of each cohort, 10 patients have stage IV NSCLC, 10 have stage III colon cancer and 10 have stage IV CRC. Prospective patients will be recruited longitudinally from January 2013 and retrospective patients are recorded longitudinally backward in time from December 2012. Both groups are patients of Medical Oncology Service of Hospital General Universitario de Elche, and both groups sign an informed consent form.

A CGA is performed in the experimental group after the first visit with oncologist and prior to therapeutic decision. This CGA includes:

* Nutritional Assessment: Mini Nutritional Assessment (MNA)
* Functional Assessment: Get up and Go, Activities of Daily Living (ADL), Instrumental Activities of Daily Living (IADL), Karnofsky Scale, Walking one Block, Number of Falls in last 6 months and Hearing Loss.
* Cognitive Assessment: Mini-Mental State Examination (MMSE-30)
* Psychological status: Geriatric Depression Scale (GDS)
* Social Support: Medical Outcomes Study Social Support Survey (MOS-SSS)
* Comorbidity and Severity of Comorbidities: Charlson Comorbidity Index and Adult Comorbidity Evaluation (ACE-27)

The evaluation includes too age, haemoglobin, Creatinine Clearance (CrCl) and presence of geriatric syndromes.

The results of this evaluation allow to calculate:

* Early mortality risk according to Soubeyran et al (JCO 2012, 30: 1829-1834) (MNA and Get up and Go):
* risk of early mortality
* no risk of early mortality.
* Toxicity to chemotherapy according to Hurria et al. (J Clin Oncol 2011, 29: 3457-3465) (age, type of cancer, dose and number of chemotherapy drugs, haemoglobin, CrCl, hearing loss, number of falls in last 6 months, ability to take medication without help (IADL), walking one block and social support (MOS-SSS):
* low risk
* medium risk
* high risk.
* Frailty group according Köhne et al (The Oncologist 2008, 13: 390-402) (ADL, IADL, comorbidity and severity of comorbidities and presence of geriatric syndromes). This information dictates the therapeutic strategy for each experimental patient:
* Group 1: standard treatment.
* Group 2: modified treatment
* Group 3: no treatment

Experimental patients will be followed for six months from CGA and their toxicity and its severity, occurrence of treatment modifications, number of hospitalizations and reasons for hospitalizations and mortality and reason of mortality will be compared with the same items of historic controls, followed too for six months from the moment the physician made the therapeutic decision.

Other data to record for both groups: sex, age, origin, leucocytes, platelets, LDH, albumin, CEA, Cr Cl, haemoglobin, subjective weight loss, corporal mass index, comorbidities, primary tumor: stage, metastases location, treatment intent: adjuvant, palliative, number of drugs, number of concomitant medications, PS according to ECOG and Karnofsky (some data are expected to be missing for historic group).

Only for historic controls, physicians should answer one question : In wich category would include the treatment recommendation? according to Köhne, The Oncologist 2008: Balducci, The Oncologist 2000; J Clin Oncol 2012:

* standard treatment
* modified treatment
* no treatment despite treatment is recommended
* no treatment

Only for historic controls two more questions should be answered:

* Has a Geriatric Evaluation been performed? Yes or No
* What sort of evaluation?

The trial records too how long does it take each test and how long does it take to complete CGA.

All information is recorded in a database with anonymous code for each subject.

Statistical analysis will consist of a descriptive analysis of sociodemographic and clinical characteristics of both cohorts. It will be performed also non-parametric analysis comparing this characteristics between the experimental groups. A descriptive analysis of daily life characteristics in experimental group will be performed, and also a non-parametric analysis comparing these variables between the experimental groups.

Changes due to CGA incorporation will be evaluated and the variables measuring the toxicity and early mortality should be correlated to the coincidence or not of the treatment performed with the one concluded by the geriatric evaluation.

Contribution of the different elements of CGA will be evaluated. A multiple regression will be performed in order to carry out an evaluation of the degree of contribution of each of the elements of the CGA.

A significance "p" less than 0.05 will be considered significant.

There are some study limitations: size, missing data for historic patients, monocentric study.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 70 years
* Outpatients
* Patients diagnosed with stage III colon cancer, stage IV colorectal cancer or stage IV NSCLC
* No previous diagnosis of cancer.
* No previous chemotherapy for current diagnosis of cancer
* Signed informed consent

Exclusion Criteria:

* Not fulfilling inclusion criteria

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2014-07-30 (Actual); Study Completion 2015-01-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAE v4.0 | 6 months
  Evaluate occurrence of toxicity in both groups, experimental and control

SECONDARY OUTCOMES:
Number of participants with occurrence of early mortality | 6 months
  Evaluate occurrence of early mortality in both groups, experimental and control
Number of Hospitalizations | 6 months
  Evaluate occurrence of hospitalizations in both groups, experimental and control
Number of participants with changes in cancer treatment related to toxicity | 6 months
  Evaluate changes in treatment in both groups, experimental and control
Number of participants with a change in therapeutic decision related to CGA | 6 months
  Evaluate impact in the treatment for cancer in elderly population with NSCLC stage IV, colon cancer stage III and CRC stage IV of a CGA
Contribution of different components of CGA to the management fo cancer | 6 months
  Analysis of the weight of ech component through multiple regression
Impact of CGA in health care in terms of human recourses and time consumption | Baseline
  Cost of CGA measured in minutes for each component of CGA and person
Predictive factors of events related to treatment | 6 months
  To detect wich conditions predispose to adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Javier Gallego, PhD, Principal Investigator — HOSPITAL GENERAL UNIVERSITARIO DE ELCHE

IPD SHARING:
Plan to Share IPD: No